CLINICAL TRIAL: NCT00829348
Title: Short Massages Service (SMS) Impact on Patient Compliance Receiving Long Term Lipid Lowering Therapy With Statins.
Brief Title: Short Message Service (SMS) Impact on Patient Compliance Receiving Long Term Lipid Lowering Therapy With Statins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Avraham Shotan, MD, Hillel Yaffe medical center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 61-2005-CTIL
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2009-12

CONDITIONS: Dyslipidemia
Keywords: Compliance; Chronic; Pharmacotherapy; Statins
MeSH Terms: conditions — Dyslipidemias; Patient Compliance; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Statins, counseling (No Intervention): 60 patients post ACS receiving the study medication + doctor/pharmacist explanation at discharge - control group
  Interventions: Other: No intervention
- Statins, Counselling, SMS (Experimental): 60 patients post ACS receiving the study medication + doctor/pharmacist explanation at discharge + daily SMS reminder service (8 PM) - study group
  Interventions: Behavioral: Short Message Service (SMS)

INTERVENTIONS:
Other: No intervention — 60 patients post ACS receiving the study medication + doctor/pharmacist explanation at discharge - control group
  Arms: Statins, counseling
Behavioral: Short Message Service (SMS) — 60 patients post ACS receiving the study medication + doctor/pharmacist explanation at discharge + daily SMS reminder service (8 PM) - study group
  Arms: Statins, Counselling, SMS

SUMMARY:
The objective of the study is to determine whether short text massages could be used successfully as a compliance aid and improve clinical outcomes in long term lipid lowering therapy.

DETAILED DESCRIPTION:
Indication: Patients discharged from the Intensive Cardiac Care Unit or the Internal Medicine Department following acute coronary syndrome (ACS) events such as unstable angina or acute myocardial infarction who will be prescribed a statin for the first time for preventing further coronary episodes.

Drug(s) and Dose/Regimen: Regular or aggressive Simvastatin therapy (dose will be adjusted according to LDL and Total Cholesterol levels). Treatment period 6 months.

Objectives: To determine whether using SMS technology can improve compliance and hence clinical outcomes in patients with long-term lipid lowering therapy.

Primary outcome: number of patients who achieve target LDL goals. Secondary outcomes: reductions of total cholesterol, LDL, LDL/HDL and CRP; increase of HDL; Readmissions due to ACS.

Study Background/Rationale/Purpose: Long-term lipid lowering therapy is the cornerstone of preventing recurrent cardiac events in patients that have experienced such episodes. Numerous studies have demonstrated the efficacy of statins in the treatment of hyperlipidemia and reduction of total mortality, vascular mortality and coronary adverse events1.

One of the main concerns affecting the success of long-term chronic drug treatments is patients' compliance and adherence to the prescribed regimen. Till date there is no gold standard system that will assure complete patient compliance.

It has been suggested to explore the possibility of using short messages service (SMS) technology to improve patients' compliance 2-18. Such technology may be effective in targeting this problem; however, no controlled trials have been conducted to validate this method in long-term lipid lowering treatments. Furthermore, Israel is one of the leading countries in terms of expansion of the mobile phone services market, making SMS a feasible and effective form of communication with patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from the Intensive Cardiac Care Unit or the Internal Medicine Department following ACS who will be prescribed a statin for the first time for preventing further coronary episodes.
* Patients in the ages of 18-80.
* Patients who own mobile phone and are familiar with SMS technology and are able to read Hebrew text.

Exclusion Criteria:

* Contra indication to study medication: active liver disease or elevated liver enzymes; hypersensitivity to Simvastatin; pregnancy and lactation.

Developed Myopathy/Rhabodmyalisis during study period.

* Developed increase in transaminases greater than 3 times the upper limit of normal.
* Current lipid lowering treatment (statins or other).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Number of patients who achieve target goals | Every three months at one year period

SECONDARY OUTCOMES:
Total cholesterol, LDL, HDL, TG | Every three months at one year period

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Shotan, MD, Study Chair — Hillel Yaffe medical center, Hadera, Israel
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel

REFERENCES:
- [Background] Consoli SM, Bruckert E, Marcantoni JP, Clavel T. [Factors associated with the opinion of hypercholesterolemic patients on the duration of their treatment. Results of the FRACTION study]. Presse Med. 2002 Sep 7;31(28):1302-8. French. PMID 12355991
- [Background] Ostojic V, Cvoriscec B, Ostojic SB, Reznikoff D, Stipic-Markovic A, Tudjman Z. Improving asthma control through telemedicine: a study of short-message service. Telemed J E Health. 2005 Feb;11(1):28-35. doi: 10.1089/tmj.2005.11.28. PMID 15785218
- [Background] Anhoj J, Moldrup C. Feasibility of collecting diary data from asthma patients through mobile phones and SMS (short message service): response rate analysis and focus group evaluation from a pilot study. J Med Internet Res. 2004 Dec 2;6(4):e42. doi: 10.2196/jmir.6.4.e42. PMID 15631966
- [Background] Vilella A, Bayas JM, Diaz MT, Guinovart C, Diez C, Simo D, Munoz A, Cerezo J. The role of mobile phones in improving vaccination rates in travelers. Prev Med. 2004 Apr;38(4):503-9. doi: 10.1016/j.ypmed.2003.12.005. PMID 15020186
- [Background] Bos A, Hoogstraten J, Prahl-Andersen B. Failed appointments in an orthodontic clinic. Am J Orthod Dentofacial Orthop. 2005 Mar;127(3):355-7. doi: 10.1016/j.ajodo.2004.11.014. PMID 15775951
- [Background] Kwon HS, Cho JH, Kim HS, Lee JH, Song BR, Oh JA, Han JH, Kim HS, Cha BY, Lee KW, Son HY, Kang SK, Lee WC, Yoon KH. Development of web-based diabetic patient management system using short message service (SMS). Diabetes Res Clin Pract. 2004 Dec;66 Suppl 1:S133-7. doi: 10.1016/j.diabres.2003.10.028. PMID 15563964
- [Background] Ferrer-Roca O, Cardenas A, Diaz-Cardama A, Pulido P. Mobile phone text messaging in the management of diabetes. J Telemed Telecare. 2004;10(5):282-5. doi: 10.1258/1357633042026341. PMID 15494086
- [Background] Power MR, Power D. Everyone here speaks TXT: deaf people using SMS in Australia and the rest of the world. J Deaf Stud Deaf Educ. 2004 Summer;9(3):333-43. doi: 10.1093/deafed/enh042. PMID 15304436
- [Background] Sherry E, Colloridi B, Warnke PH. Short message service (SMS): a useful communication tool for surgeons. ANZ J Surg. 2002 May;72(5):369. doi: 10.1046/j.1445-2197.2002.02411.x. No abstract available. PMID 14696592
- [Background] Marquez Contreras E, de la Figuera von Wichmann M, Gil Guillen V, Ylla-Catala A, Figueras M, Balana M, Naval J. [Effectiveness of an intervention to provide information to patients with hypertension as short text messages and reminders sent to their mobile phone (HTA-Alert)]. Aten Primaria. 2004 Nov 15;34(8):399-405. doi: 10.1016/s0212-6567(04)78922-2. Spanish. PMID 15546536
- [Background] Neville R, Greene A, McLeod J, Tracey A, Surie J. Mobile phone text messaging can help young people manage asthma. BMJ. 2002 Sep 14;325(7364):600. doi: 10.1136/bmj.325.7364.600/a. No abstract available. PMID 12228151
- [Background] Bramley D, Riddell T, Whittaker R, Corbett T, Lin RB, Wills M, Jones M, Rodgers A. Smoking cessation using mobile phone text messaging is as effective in Maori as non-Maori. N Z Med J. 2005 Jun 3;118(1216):U1494. PMID 15937529
- [Background] Lieu TA, Capra AM, Makol J, Black SB, Shinefield HR. Effectiveness and cost-effectiveness of letters, automated telephone messages, or both for underimmunized children in a health maintenance organization. Pediatrics. 1998 Apr;101(4):E3. doi: 10.1542/peds.101.4.e3. PMID 9521970
- [Background] Obermayer JL, Riley WT, Asif O, Jean-Mary J. College smoking-cessation using cell phone text messaging. J Am Coll Health. 2004 Sep-Oct;53(2):71-8. doi: 10.3200/JACH.53.2.71-78. PMID 15495883
- [Background] Dyer O. Patients will be reminded of appointments by text messages. BMJ. 2003 Jun 14;326(7402):1281. doi: 10.1136/bmj.326.7402.1281-a. No abstract available. PMID 12805131
- [Background] Lauruska V, Kubilinskas E. A system for teleconsulting, communication and distance learning for people with disabilities. J Telemed Telecare. 2002;8 Suppl 2:49-50. doi: 10.1177/1357633X020080S222. PMID 12217133
- [Background] Ferrer-Roca O, Franco Burbano K, Cardenas A, Pulido P, Diaz-Cardama A. Web-based diabetes control. J Telemed Telecare. 2004;10(5):277-81. doi: 10.1258/1357633042026288. PMID 15494085